CLINICAL TRIAL: NCT01501604
Title: An Open Label, Phase II Trial of BKM120 in Cancers With PIK3CA Activating Mutations
Brief Title: BKM120 in Cancers With PIK3CA Activating Mutations
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study has been closed due to lack of accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Jeffrey Engelman, Director, Thoracic Oncology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-211
Record Dates: First submitted 2011-12-27; First posted 2011-12-29 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Lung Cancer; Breast Cancer; Colorectal Cancer; Cholangiocarcinoma; Solid Tumors
Keywords: PIK3CA mutation; Advanced solid tumors
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Cholangiocarcinoma | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: BKM120 — 100 MG PO QD in cycles of 28 days

SUMMARY:
In people whos cancers have a PIK3CA mutation, this trial will be evaluating the drug BKM120 as a possible treatment. BKM120 works by blocking the phosphatidylinositol-3-kinase (PI3K)pathway, thereby inhibiting tumor growth and survival.

The purpose of this study is to learn if the study drug BKM120 can shrink or slow the growth of your tumor. The safety of BKM120 will also be studied. Your physical state, symptoms, change in the size of your tumor, and laboratory findings obtained while you are on study will help the research team decide if BKM120 is safe and effective in patients with advanced cancers.

DETAILED DESCRIPTION:
Subjects enrolled in this study will receive BKM120 once daily, orally, in cycles of 28 days.

During Cycles 1 and 2, the following tests and procedures will be done on days 1 and 15:

* physical exam
* performance status
* blood tests
* pregnancy test (if applicable)
* neuropsychiatric assessments

Starting at Cycle 2 and then every other cycle thereafter (approximately every 8 weeks) tumor assessment will be performed by CT/MRI or PET scan. A chest x-ray will also be performed every 8 weeks.

Beginning with Cycle 3, the following tests/procedures will be performed on Day 1 of each cycle:

* physical exam
* performance status
* blood tests
* neuropsychiatric assessments

ELIGIBILITY:
Inclusion Criteria:

* At least 1 site of measurable disease
* Life expectancy >/= 12 weeks
* Adequate marrow and organ function
* Diagnosis of lung cancer, breast cancer, colorectal cancer, cholangiocarcinoma, gastric cancer, pancreatic cancer, prostate cancer, uterine cancer, ovarian cancer, esophageal cancer, or head and neck cancer
* Pathologically documented, definitively diagnosed, advanced solid tuor that is refractory to standard treatment, for which no standard therapy is available, or the subject refuses standard therapy
* Cancer must have at least one of the following PIK3CA mutations: E542K, E545K, H1047R, H1047L. The PIK3CA mutation must be documented in a CLIA approved laboratory

Exclusion Criteria:

* Prior treatment with a P13K inhibitor
* Known hypersensitivity to BKM120 or its excipients
* Untreated brain metastases
* Acute or chronic liver, renal disease or pancreatitis
* Currently treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A
* Diarrhea >/= CTCAE grade 2
* Any concurrent severe and/or uncontrolled medical condition
* Active cardiac disease
* History of cardiac dysfunction
* Poorly controlled diabetes mellitus or steroid-induced diabetes mellitus
* Significant symptomatic deterioration of lung function
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKDM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant
* Pregnant or breast-feeding
* Known diagnosis of HIV infection
* History of another malignancy within 3 years, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix
* Unable to swallow the medication in its prescribed form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Response Rate | 2 years
  Objective Response Rate (CR or PR) by RECIST 1.1 criteria

SECONDARY OUTCOMES:
Clinical Benefit Rate | 2 years
  Clinical Benefit Rate (CR, PR, or SD) by RECIST 1.1 criteria
Survival | 2 years
  Progression Free Survival (PFS)
Clinical Benefit | 2 years
  Determine if the presence of specific co-existing mutations may influence clinical benefit from BKM120

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Engelman, MD, PhD, Principal Investigator — Massachusetts General Hospital